CLINICAL TRIAL: NCT03640338
Title: The Efficacy of Continuous Cold-Therapy on Postoperative Pain and Narcotics Use Following Spinal Fusion
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Limiting funding sources forced us to withdraw the study.
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 18050401
Record Dates: First submitted 2018-08-03; First posted 2018-08-21 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Radiculopathy; Central Spinal Stenosis; Foraminal Stenosis; Herniated Nucleus Pulposus; Degenerative Disc Disease; Isthmic Spondylolisthesis; Degenerative Spondylolisthesis
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold-therapy system (Experimental): Patients will receive a cold-therapy system postoperatively (Polar Care Kodiak, Breg®) and will use the system during inpatient stay and during the first 14 days post-discharge.
  Interventions: Device: Cold-Therapy System
- Standard care (ice-pack) (No Intervention): Patients will use disposable ice-pack as per standard of care

INTERVENTIONS:
Device: Cold-Therapy System — After surgery, participants assigned to this group will receive the cold-therapy system to use at the hospital and during the first 2 weeks following discharge.
  Other Names: Polar Care Kodiak, Breg®
  Arms: Cold-therapy system

SUMMARY:
Patient outcomes and satisfaction are an ever-increasing priority in surgical specialties. Cryotherapy has been utilized following spine surgery as an adjunct therapy to reduce postoperative inflammation and improve patient outcomes. However, limited studies have investigated the effect of cryotherapy on postoperative pain and narcotics use. Fountas et al. performed a randomized controlled trial to assess the impact of postoperative cryotherapy following single-level lumbar microdiscectomy. The authors reported patients receiving cryotherapy required significantly less pain medication (0.058 mg/kg/hr versus 0.067 mg/kg/hr, p<0.001) and had shorter hospital stays (1.71 days versus 2.65 days, p<0.001) as compared to the control group. In another randomized trial of single-level lumbar discectomy patients, Murata et al. demonstrated cryotherapy to have no significant effect on VAS inpatient pain scores or postoperative blood loss.

DETAILED DESCRIPTION:
The purpose of this study is to determine if postoperative cryotherapy with a cold-therapy system reduces postoperative pain and narcotic consumption following single and multi-level spinal fusion.

The investigators hypothesize that patients undergoing lumbar spinal fusion who receive postoperative cryotherapy treatment with a cold-therapy system will have reduced inpatient pain scores and require less narcotics as compared to patients that receive standard care (ice pack).

ELIGIBILITY:
Inclusion Criteria:

1. Single or multi-level lumbar spinal fusion for degenerative pathology, including: radiculopathy, central spinal stenosis, foraminal stenosis, herniated nucleus pulposus, degenerative disc disease, and isthmic or degenerative spondylolisthesis.
2. Patient able to provide informed consent

Exclusion Criteria:

1. Chronic preoperative narcotic use defined as daily narcotic use for the past 6 months prior to surgery
2. Workers' compensation insurance claim
3. Active or history of malignancy
4. Unable to speak, read, or comprehend English language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | 2 year postoperative
  Average daily Visual Analog Scale (VAS) survey, which measures pain, for the duration of hospital stay and postoperative VAS scores will be recorded for 2 years postoperatively. This information will be collected through a survey that will be administered upon patient discharge. Patients will be asked to return the completed survey to the research team.
  VAS scale ranges from 0 - 100 mm, with 100 representing maximum pain and 0 representing no pain.
Narcotics Consumption | 2 weeks postoperative
  Total, daily, and hourly narcotics consumption during the hospitalization. Narcotic consumption will be recorded for 2 weeks following discharge. Patients will be asked to report the number of narcotic pills taken each day. This information will be collected through a survey that will be administered upon patient discharge. Patients will be asked to return the completed survey to the research team.

SECONDARY OUTCOMES:
Bony fusion | 2 year postoperative
  Postoperative radiographs and CT scan will be used to assess fusion.
Disability | 2 year postoperative
  Postoperative Oswestry Disability Index (ODI) survey scores will be compared to preoperative values.
  ODI measures disability for lumbar patients. The scale ranges from 0% to 100%. 0-20% represents minimal disability, 21-40% represents moderate disability, 41-60% represents severe disability, 61%-80% represents a crippled state, and 81-100% represents a bed-bound patient.
Physical Function: Patient-Reported Outcomes Measurement Information System (PROMIS) | 2 year postoperative
  Postoperative PROMIS scores will be compared to preoperative values.
  PROMIS evaluates physical function through a series of questions covering level of difficulty with normal daily activities. A score of 5 represents "without any difficulty" and a score of 1 represents "unable to do".
General Health Status: Short-Form (SF-12) | 2 year postoperative
  Postoperative SF-12 scores will be compared to preoperative values.
  SF-12 evaluates the general health status of the patient. A minimum score of 0 represents the lowest level of health, while a maximum score of 100 represents the highest level of health.
Length of Stay | Up to 2 weeks
  The number of hours of hospitalization from entering the recovery room (time zero) until patient meets discharge criteria.
Disposition on discharge | Up to 2 weeks
  This outcome evaluates where the patient will return to after their inpatient stay. This could include, but is not limited to, their home, a rehabilitation facility, or a skilled nursing facility.

CONTACTS AND LOCATIONS:
Overall Officials: Kern Singh, MD, Principal Investigator — Rush University Medical Center

IPD SHARING:
Plan to Share IPD: No